CLINICAL TRIAL: NCT05548257
Title: Mortality and Related Risk Factors After Hip Arthroplasty, a Retrospective Study
Brief Title: Mortality and Related Risk Factors After Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2022-012-B
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Fracture of Neck of Femur (Hip); Femoral Head Necrosis; Dislocation of Hip Joint; Dysplasia of Hip Joint
MeSH Terms: conditions — Femoral Neck Fractures; Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients were reviewed

SUMMARY:
The patients who underwent hip arthroplasty in our hospital from January 2017 to December 2020 were reviewed. The perioperative data were collected, and then the mortality was calculated and the risk factors were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hip arthroplasty in Renji Hospital during 2017.1-2020.12

Exclusion Criteria:

* Patients who did not undergo surgery after admission Age < 18 years Patients undergoing the second operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing hip arthroplasty in Renji Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-08-04 (Estimated); Study Completion 2023-08-04 (Estimated)

PRIMARY OUTCOMES:
Risk factors of mortality one year after operation | From about even days before operation to 12 months after operation

SECONDARY OUTCOMES:
Risk factors of lower activities of daily living score at 12 months after operation | From about even days before operation to 12 months after operation

IPD SHARING:
Plan to Share IPD: Yes